CLINICAL TRIAL: NCT01097993
Title: A Single-centre, Randomised, Double-blind, Controlled, Parallel-group Study to Evaluate the Effect of a Fermented Dairy Product on Abdominal Distension, Digestive Symptoms and Rectal Sensitivity in Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NU324
Record Dates: First submitted 2010-03-29; First posted 2010-04-02 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Women With IBS-C
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Experimental)
  Interventions: Other: 1-fermented dairy product
- 2 = Control product (Active Comparator)
  Interventions: Other: 2- milk-based non-fermented dairy product (control product)

INTERVENTIONS:
Other: 1-fermented dairy product — Arm 1 - Intervention 1 (probiotics)
  Arms: 1 = Tested product
Other: 2- milk-based non-fermented dairy product (control product) — Arm 2 - Intervention 2 (control)
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to evaluate the effect of a commercially available fermented dairy product containing probiotics (4 weeks, twice a day) on abdominal distension in IBS patients with constipation (IBS-C).

ELIGIBILITY:
Inclusion Criteria:

* female
* Age: 18-70

Exclusion Criteria:

* NA

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Mean abdominal distension after a 4-week period of product consumption in IBS-C patients | 0-4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Hospital, Manchester, United Kingdom